CLINICAL TRIAL: NCT03003130
Title: A Randomized, Multi-center, Evaluator-blinded Study to Evaluate the Efficacy and Safety of Restylane Defyne Compared to Restylane for Correction of Moderate to Severe Nasolabial Folds
Brief Title: Restylane Defyne Compared to Restylane for Correction of Moderate to Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43CH1508
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2021-07

CONDITIONS: Nasolabial Folds in Chinese Population
Keywords: Hyaluronic acid; Comparative study; NLF

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restylane Defyne (Experimental): Single injection and optional touch up injection with Restylane Defyne in NLF
  Interventions: Device: Restylane Defyne
- Restylane (Active Comparator): Single injection and optional touch up injection with Restylane in NLF
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Restylane Defyne — Intradermal injection
  Arms: Restylane Defyne
Device: Restylane — Intradermal injection
  Arms: Restylane

SUMMARY:
This is a randomized, split face, multicenter study to evaluate the efficacy and safety of Restylane Defyne compared to Restylane in correction of NLFs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Men or women aged 18 years of age or older of Chinese origin.
3. Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the lower orbital rim for the duration of the study.
4. Intent to undergo correction of both NLFs with a wrinkle severity in WSRS of either 3 on both sides or 4 on both sides, as assessed by the blinded evaluator.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) Gel and/or local anesthetics, e.g., lidocaine or other amide-type anesthetics.
2. Previous tissue revitalization treatment below the level of the lower orbital rim within 6 months before treatment.
3. Previous surgery or tattoo in the area to be treated.
4. Previous tissue augmentation therapy or contouring with any permanent (nonbiodegradable) or semi-permanent facial tissue augmentation therapy or autologous fat or permanent implant below the level of the lower orbital rim.
5. Previous use of neurotoxins or any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy below the level of the lower orbital rim within 12 months before treatment.
6. Scars or deformities, active skin disease, inflammation or related conditions such as infection, perioral dermatitis, seborrheic dermatitis, eczema, rosacea, acne, psoriasis, and herpes zoster near or in the area to be treated.
7. Other condition preventing the subject from entering the study in the Investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Med AB, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject have 2 NLFs, the right/left one. According to protocol that Each subject will be randomized to one of two treatment sequences; either Restylane Defyne in the right NLF followed by Restylane in the left NLF, or Restylane in the right NLF followed by Restylane Defyne in the left NLF. Arms/Groups are combined because right/left side is not statistical factors.
Groups:
- Restylane Defyne in the Right NLF Followed by Restylane in the Left NLF: Restylane Defyne treated in the right NLF followed by Restylane in the left NLF
- Restylane in the Right NLF Followed by Restylane Defyne in the Left NLF: Restylane treated in the right NLF followed by Restylane Defyne in the left NLF
Period: Overall Study
Arm/Group | Restylane Defyne in the Right NLF Followed by Restylane in the Left NLF | Restylane in the Right NLF Followed by Restylane Defyne in the Left NLF
Started | 88 | 87
Completed | 80 | 80
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Population: Each subject will be randomized to one of two treatment sequences; either Restylane Defyne in the subject's right NLF followed by Restylane in the subject's left NLF, or Restylane in the subject's right NLF followed by Restylane Defyne in the subject's left NLF.
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Defyne in the Right NLF Followed by Restylane in the Left NLF | Restylane in the Right NLF Followed by Restylane Defyne in the Left NLF | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 86 | 174
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8.7) | 44 (8.7) | NA (NA) — This data is not applicable for study.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 83 | 166
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 88 | 87 | 175
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 88 | 87 | 175

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders, Defined by at Least 1-point Improvement From Baseline on the WSRS.
Description: The Wrinkle Severity Rating Scale (WSRS) is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds.
  Grade 1 Absent: No visible fold; continuous skin line Grade 2 Mild: Shallow but visible fold with a slight indentation; minor facial feature Implant is expected to produce a slight improvement in appearance Grade 3 Moderate: Moderately deep folds; clear facial feature visible at normal appearance but not when stretched. Excellent correction is expected from injectable implant Grade 4 Severe: Very long and deep fold; prominent facial feature; less than 2-mm visible fold when stretched Significant improvement is expected from injectable implant Grade 5 Extreme: Extremely deep and long fold; detrimental to facial appearance; 2- to 4-mm V-shaped fold when stretched. Unlikely to have satisfactory correction with injectable implant alone
Time Frame: 6 month
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Restylane Defyne in the Right NLF Followed by Restylane in the Left NLF | Restylane in the Right NLF Followed by Restylane Defyne in the Left NLF
Number analyzed (Participants) | 87 | 86
percentage of subjects | 72.9 [66.3 to 79.6] | 72.8 [66.1 to 79.5]

ADVERSE EVENTS:
Time Frame: 1 year.
Description: According to the subject's treatment randomization.Each subject should be questioned about AEs at each study visit following the screening visit. The question asked should be: "Since your last clinical visit have you had any health problems?", and or obtained from signs and symptoms from examination, lab test, self observations, diary or spontaneous reports from subject. Since each subject will receive Restylane and Restylane Defyne, then AE was collected per subject, not per intervention.
Groups:
- Restylane Defyne; Restylane: Since all participants received both Restylane and Restylane Defyne treatments, the appropriate way to present Adverse Events to include two Arms eflecting all participants who received each intervention during the study.
Arm/Group | Restylane Defyne | Restylane
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/175
Serious Adverse Events (participants affected / at risk) | 3/175 | 3/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Defyne (N=175) | Restylane (N=175)
Retinal detachment* (Eye disorders) | 1 (1) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03003130/Prot_002.pdf
  • Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT03003130/SAP_003.pdf